CLINICAL TRIAL: NCT02417324
Title: International HIT-MED Registry (I-HIT-MED) for Children, Adolescents, and Adults With Medulloblastoma, Ependymoma, Pineoblastoma, CNS-primitive Neuroectodermal Tumours
Brief Title: International HIT-MED Registry (I-HIT-MED)
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: I-HIT-MED Registry
Record Dates: First submitted 2015-02-04; First posted 2015-04-15 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Childhood Brain Tumor
Keywords: medulloblastoma; ependymoma; pineal tumour; CPT
MeSH Terms: conditions — Medulloblastoma; Ependymoma; Pinealoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tumour samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The I-HIT-MED registry registers clinical of children and adults with medulloblastoma, ependymoma, pineal tumours, or choroid plexus tumours in Germany and other countries that fulfil national ethic requirements for participation in this registry. These tumours are rare diseases, and many patients are treated outside of clinical trials. The I-HIT-MED registry allows collection of data und biological material from those patients, and provides a basis for standard treatment recommendations and counselling. It aims to improve the international cooperation and the medical knowledge in these rare diseases. Within the I-HIT-MED registry, it is a goal to maintain and improve networks for quality assurance in national groups where they are already established, and to support the implementation in national groups, where there is no quality assurance network yet.

DETAILED DESCRIPTION:
The following patients can be included in this registry:

Children and adults with

* Medulloblastoma (MB)
* Ependymoma
* Pineal Tumours
* Chroroid plexus tumours

Objectives of this registry:

To prospectively evaluate the clinical courses of patients with the eligible brain tumours, considering neuroradiological, pathological, and molecular / biological characteristics of the tumour and individual standard treatment data.

To collect biological specimens (tumour, CSF, peripheral blood) or their data to perform biological studies on

* disease aetiology
* molecular / biological risk factors influencing treatment response and survival
* potential targets for drug treatment in future patients

To assess the use of systems for quality assurance during diagnosis and treatment of brain tumours.

To assess long-term follow-up, quality of survival, neuropsychology, and other patient-centred research in these very rare tumour subtypes in the context of the registry or in cooperation with external collaborators.

ELIGIBILITY:
Inclusion Criteria:

* all patients with above mentioned diagnosis of all ages (except for ependymoma WHO I°, pineal parenchymal tumour of intermediate differentiation and papillary tumour of the pineal region, who will be registered only if primary diagnosis was before the 18th birthday)
* any localisation of the primary tumour
* all clinical stages
* First diagnosis after 01.01.2012
* No inclusion into a prospective clinical trial for the same diagnosis, due to non-eligibility, national lack of trial approval, or individual refusal of participation.
* Written informed consent for data transfer and tumour sample submission according to the laws of each participating country is necessary.
* National and/ or local ethical committee approval according to the laws of each participating country is necessary.

Exclusion Criteria:

* Registration in another clinical trial for the same diagnosis (relapse is defined as a second diagnosis).
* Lack of valid ethical committee approval.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults with
  * Medulloblastoma (MB)
  * Ependymoma
  * CNS-primitive neuroectodermal tumours (CNS-PNET) including CNS neuroblastoma, CNS ganglioneuroblastoma, Medulloepithelioma, Ependymoblastoma, CNS-PNET not otherwise specified (NOS)
  * Pineoblastoma
  * Pineal parenchymal tumour of intermediate differentiation
  * Papillary tumour of the pineal region Who are not included in prospective clinical trials for these conditions
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-01; Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 10 years
  Due to the explorative character of the registry, outcome measures are not strictly defined. We added the most common outcome measures.

SECONDARY OUTCOMES:
Pattern of relapse | 10 years
Overall survival | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Rutkowski, Prof., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (57):
- Germany (57):
  - University Hospital Aachen, Aachen
  - Klinikum Augsburg, Augsburg
  - Helios Klinikum Berlin-Buch, Berlin
  - Charite Campus, University of Berlin, Berlin
  - Evangelisches Krankenhaus Bielefeld, Bielefeld
  - Klinikum Braunschweig, Braunschweig
  - Klinikum Bremen-Mitte, Bremen
  - Klinikum Chemnitz, Chemnitz
  - University Hospital Cologne, Cologne
  - Carl-Thiem-Klinikum Cottbus, Cottbus
  - Vestische Kinder- und Jugendklinik, University Witten/Herdecke, Datteln
  - Klinikum Dortmund, Dortmund
  - University Hospital Dresden, Dresden
  - Klinikum Duisburg, Duisburg
  - Universitäts-Kinderklinik Düsseldorf, Düsseldorf
  - HELIOS Klinikum-Erfurt, Erfurt
  - University Hospital Erlangen, Erlangen
  - University Hospital Essen, Essen
  - University Hospital Frankfurt/Main, Frankfurt
  - University Hospital Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Gießen und Marburg, Giessen
  - Georg-August-Universität Göttingen, Göttingen
  - University Hospital Greifswald, Greifswald
  - University Hospital Halle/Saale, Halle
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Angelika-Lautenschläger-Klinik, Heidelberg
  - SLK-Kliniken, Heilbronn
  - Gemeinschaftskrankenhaus Herdecke, Herdecke
  - University Hospital Homburg/Saar, Homburg
  - University Hopsital Jena, Jena
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Klinikum Kassel, Kassel
  - UK-SH Campus Kiel, Kiel
  - Gemeinschaftsklinikum Koblenz-Mayen, Koblenz
  - HELIOS Klinikum Krefeld, Krefeld
  - University Hospital Leipzig, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - University Hospital Magdeburg, Magdeburg
  - University Hospital Mainz, Mainz
  - University Hospital Mannheim, Mannheim
  - Johannes Wesling Klinikum Minden, Minden
  - Universität München - von Haunersches, München
  - Klinikum Schwabing, Pediatric Hospital of Technical University, München
  - Universitätsklinikum Münster, Münster
  - Cnopf'sche Kinderklinik, Nuremberg
  - Klinikum Oldenburg, Oldenburg
  - University Hospital Regensburg, Regensburg
  - University Hospital Rostock, Rostock
  - Asklepios Klinik Sankt Augustin, Sankt Augustin
  - Helios Kliniken Schwerin, Schwerin
  - Klinikum Stuttgart, Stuttgart
  - Universitätsklinik Tübingen, Tübingen
  - University Hospital Ulm, Ulm
  - Dr. Horst Schmidt Kliniken, Wiesbaden
  - Klinikum der Stadt Wolfsburg, Wolfsburg
  - Universotätsklinikum Würzburg, Würzburg